CLINICAL TRIAL: NCT06359184
Title: Examining the Effect of Yoga on Maternal Stress and Sleep Quality of Mother and Baby, Mother's Feeding Attitude and Baby's Feeding Behavior: Randomized Controlled Study.
Brief Title: Yoga, Mother's Stress and Baby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe Nur Ozan, occupational therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO21/1011
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Mother-Child Relations
Keywords: yoga; mothers; baby; stress; sleep; nutrition
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga (Experimental): Yoga will be practiced 1 hour a day, 2 days a week for 8 weeks, for a total of 16 hours.
  Interventions: Other: yoga
- control (Placebo Comparator): No intervention is applied for 8 weeks.
  Interventions: Other: control

INTERVENTIONS:
Other: yoga — 1 hour yoga practice 2 days a week for 8 weeks
  Arms: yoga
Other: control — no intervention for 8 weeks
  Arms: control

SUMMARY:
The aim of this study is to examine the effects of yoga on the stress of mothers with babies with sleep and feeding problems, the mother-infant relationship, and the sleep and nutrition of the mother and the baby. 55 mothers with babies with sleep and feeding problems were included in the study. Mothers were randomly divided into two groups: yoga (n=29) and control group (n=26). Yoga training was applied to 29 mothers in the study group via video conferencing, 2 days a week, 1 hour a day for 8 weeks, while the mothers in the control group were given second evaluations 8 weeks after the first evaluation, without any intervention. Mothers were evaluated with the Perceived Stress Scale (PSS) for stress levels, with Parent-Child Containing Function Scale for the mother-infant relationship, with the Infancy and Early Childhood Feeding Process Mother'sAttitudes Scale for their attitudes towards the feeding process of their babies, and with Attitude Scale for Healthy Nutrition (ASHN) for their own nutrition attitudes, with Pittsburg Sleep Quality (PSQI) for sleep quality and babies with Infancy Period Adaptive Eating Behavior Scale for feeding problems, with Brief Infant/Child Sleep Questionnaire (BISQ) for sleep problems.

ELIGIBILITY:
Inclusion Criteria:

Parents living together The child must have at least one of the 3 problems listed below on the Infant/Child Sleep Problem Brief Diagnostic Form.

1. Waking up more than three times a night
2. Waking up at night and being sleepless for more than 1 hour
3. Total sleep time is less than 9 hours Having a score above 25 on the Infancy Adaptive Eating Behavior Scale

Exclusion Criteria:

The child has any developmental, neurological, orthopedic and/or psychiatric diagnosis Presence of a condition that prevents the mother from exercising (neurological, cardiovascular, orthopedic, etc.)

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | At the beginning and end of 8 weeks
  Evaluated for mother's stress level. It evaluates the participants on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4).
Infancy and Early Childhood Feeding Process Mother's Attitudes Scale | At the beginning and end of 8 weeks
  Evaluated Mother's attitudes towards the feeding process of their babies
Pittsburg Sleep Quality (PSQI) | At the beginning and end of 8 weeks
  Evaluated mother's sleep quality
Period Adaptive Eating Behavior Scale | At the beginning and end of 8 weeks
  Evaluated babies feeding problems
Brief Infant/Child Sleep Questionnaire (BISQ) | At the beginning and end of 8 weeks
  Evaluated babies sleep problems. If at least one of the following three conditions occurs, it is determined that the baby/child has a sleep problem; 1) The baby/child wakes up more than three times a night, 2) The baby/child wakes up at night and remains sleepless for more than an hour, or, 3) The baby/child's total sleep time is less than 9 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayşe Nur Ozan, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No